CLINICAL TRIAL: NCT07259070
Title: Multicenter, Single-Arm Exploratory Phase I Clinical Study on the Safety and Efficacy of Fully Human BAFF-R Chimeric Antigen Receptor T-Cell Injection in Participants With Relapsed/Refractory BAFF-R-Positive B-Cell Lymphoma
Brief Title: Multicenter, Single-Arm Exploratory Phase I Clinical Study (Assessment of Safety and Efficacy) of Fully Human BAFF-R Chimeric Antigen Receptor T-Cell Injection in Relapsed/Refractory BAFF-R-Positive B-Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025018
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: DLBCL; CLL; FL; MCL; WM; MZL

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAFF-R CAR-T for the Treatment of Relapsed and Refractory BAFF-R-Positive B-Cell Lymphoma (Other)
  Interventions: Drug: BAFF-R CAR-T

INTERVENTIONS:
Drug: BAFF-R CAR-T — Eligible participants should receive preconditioning 5 to 3 days prior to CAR-T cell infusion. The recommended preconditioning regimen is fludarabine (30 mg/m²/day for 3 days) and cyclophosphamide (300 mg/m²/day for 3 days) (Flu/Cy).
  Thirty minutes before the infusion, medications for preventing allergic reactions should be administered: 25 mg of promethazine hydrochloride or 12.5 mg of diphenhydramine, which can be given via intramuscular injection or oral administration.
  In Phase1 bispecific maintenance therapy will be divided into three dose groups, using a "3 + 3" dose escalation design. In Phase 2, the Maximum Tolerated Dose (MTD) identified in Phase 1 will be used, and the study will be expanded to enroll 20 participants.

SUMMARY:
The aim of this study is to analyze the safety of BAFF-R Chimeric Antigen Receptor T-Cell Injection (BAFF-R CAR-T) in participants with relapsed/refractory BAFF-R-positive B-cell lymphoma and explore the Maximum Tolerated Dose (MTD).

The secondary objective of this study is to explore the efficacy of BAFF-R CAR-T in participants with relapsed/refractory BAFF-R-positive B-cell lymphoma.

The study also aims to explore the pharmacokinetic characteristics of BAFF-R CAR-T in vivo and the impact of BAFF-R CAR-T on lymphocyte subsets in vivo.

DETAILED DESCRIPTION:
This is an investigator-initiated dose-escalation clinical study. Its primary objectives are to evaluate the safety of BAFF-R CAR-T in participants with relapsed/refractory BAFF-R-positive B-cell lymphoma and explore the Maximum Tolerated Dose (MTD) of BAFF-R CAR-T for this patient population. Additionally, the study will investigate the efficacy and pharmacokinetic characteristics of BAFF-R CAR-T in these participants.

To evaluate the safety and preliminary dose range of BAFF-R CAR-T in participants with relapsed/refractory BAFF-R-positive B-cell lymphoma, the dose groups of this trial are as follows:Dose Group 1: 1 × 10⁶ CAR⁺ T Cells/kg, Dose Group 2: 2 × 10⁶ CAR⁺ T Cells/kg, Dose Group 3: 3 × 10⁶ CAR⁺ T Cells/kg.The dose design of this study refers to the "3+3" dose escalation design for the first-in-human (FIH) trial of new drugs.

For each dose group, there must be a 14-day interval after the first participant completes BAFF-R CAR-T infusion before subsequent participants can receive BAFF-R CAR-T infusion.

If 2 cases of Dose-Limiting Toxicity (DLT) occur in the Dose 1 group, the investigators will decide whether to explore a lower dose group.

After the completion of the dose escalation phase, a decision on whether to proceed with the dose expansion phase and the determination of the dose for this phase will be made based on safety and Pharmacokinetic (PK) data.

In the dose expansion phase, after the completion of the dose escalation phase, the investigators will first identify the optimal dose group based on the available data, including preliminary efficacy and/or PK data. Subsequently, additional participants may be enrolled to receive cell infusion until the sample size reaches 20 cases. This is to further evaluate the tolerability, safety, and efficacy of the BAFF-R CAR-T cell injection.

The study process includes the screening period, apheresis period, baseline and chemotherapy preconditioning period, BAFF-R CAR-T infusion period, and post-infusion follow-up period for safety and efficacy.

After signing the Informed Consent Form (ICF), participants undergo screening examinations. Those who meet the enrollment criteria receive peripheral blood mononuclear cell (PBMC) apheresis, which is used for BAFF-R CAR-T preparation. The cell preparation takes 15 to 25 days. Participants receive lymphodepleting preconditioning 4 to 2 days before BAFF-R CAR-T infusion (Day 0) and complete the baseline assessment. BAFF-R CAR-T is administered via intravenous infusion as a single dose. After BAFF-R CAR-T infusion, follow-up for safety and efficacy is conducted. The follow-up content includes physical examinations, vital signs monitoring, laboratory tests, imaging examinations, and treatment efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

1.Relapsed and refractory (R/R) BAFF-R-positive B-cell lymphoma:The diagnosis of B-cell lymphoma must be confirmed in accordance with the NCCN Clinical Practice Guidelines in Oncology: B-Cell Lymphomas (Version 1.2020) (NCCN: National Comprehensive Cancer Network).The expression of BAFF-R on tumor cells must be detected by flow cytometry (for patients where current clinical sampling is not feasible, test results obtained within 90 days prior to signing the informed consent form are acceptable). Investigators will determine whether to accept test results from external hospitals and whether the patient is eligible for enrollment.In accordance with the 2014 Lugano Classification, B-cell lymphoma patients must have at least one measurable lesion with a longest diameter ≥ 1.5 cm, or bone marrow involvement confirmed by bone marrow flow cytometry.Patients who have received CD19-targeted therapy are also eligible for enrollment, including those who have undergone:

1. :Relapsed and refractory (R/R) mantle cell lymphoma (MCL):Histologically confirmed MCL;Relapsed or refractory after at least 2 lines of prior treatment (including anti-CD20 monoclonal antibody and Bruton's tyrosine kinase inhibitor [BTKi]).
2. :Relapsed and refractory (R/R) chronic lymphocytic leukemia (CLL):Histologically confirmed CLL;Patients who have received at least immunochemotherapy and are refractory to both BTK inhibitors and B-cell lymphoma 2 (BCL2) inhibitors.
3. :Relapsed and refractory (R/R) diffuse large B-cell lymphoma (DLBCL):Histologically confirmed DLBCL;Patients who have received anthracycline-based therapy and anti-CD20 monoclonal antibody therapy, and have undergone at least 2 lines of treatment in total; or patients who failed to achieve remission, progressed, or relapsed within 12 months after initial standard treatment.
4. :Relapsed and refractory (R/R) follicular lymphoma (FL):Histologically confirmed FL (Grade 1-3a);Patients who have received anti-CD20 monoclonal antibody-containing therapy and have undergone at least 2 lines of treatment in total; or patients who relapsed within 24 months after initial treatment.
5. :Relapsed and refractory (R/R) marginal zone lymphoma (MZL):Histologically confirmed MZL;Patients who have received anti-CD20 monoclonal antibody-containing therapy, have undergone at least 2 lines of treatment in total and relapsed thereafter; or patients who relapsed within 24 months after initial treatment.
6. :Relapsed and refractory (R/R) Waldenström macroglobulinemia (WM):Histologically confirmed WM;Patients who have received anti-CD20 monoclonal antibody-containing therapy and BTK inhibitor-containing therapy (among other medications), and have undergone at least 2 lines of treatment in total; or patients who relapsed within 24 months after initial treatment.

2.Aged ≥ 18 years and ≤ 75 years, with no restriction on gender. 3.Expected survival time ≥ 12 weeks. 4.Serum total bilirubin ≤ 37.2 μmol/L (for patients with Gilbert syndrome: serum total bilirubin ≤ 3.0 × upper limit of normal [ULN], direct bilirubin ≤ 1.5 × ULN); estimated glomerular filtration rate [eGFR] (calculated by CKD-EPI formula) ≥ 30 ml/min/1.73m²; alanine aminotransferase [ALT] and aspartate aminotransferase [AST] < 2.5 × upper limit of normal [ULN].

5.Eastern Cooperative Oncology Group (ECOG) performance status of 0-1. 6.Left ventricular ejection fraction (LVEF) ≥ 50% as diagnosed by echocardiography; oxygen saturation > 91%.

7.The participant and their spouse/partner must agree to use effective barrier or pharmaceutical contraceptive methods from the time the participant signs the informed consent form until one year after CAR-T cell infusion. For female participants of childbearing potential, serum or urine pregnancy test results must be negative during the screening period.

8.Voluntarily participate in this trial and sign the Informed Consent Form (ICF).

1. ： The patient has a full understanding of this study, voluntarily agrees to participate, and signs the Informed Consent Form (ICF).
2. ：Aged ≥ 18 years and ≤ 75 years, with no restriction on gender.

Exclusion Criteria:

1. Patients with a history of allergy to any component of the cellular product.
2. Patients with acute graft-versus-host disease (aGVHD) graded as Grade II-IV according to the Glucksberg criteria, or with severity graded as Grade B-D according to the IBMTR index; patients with acute or chronic graft-versus-host disease (cGVHD) requiring systemic treatment within 4 weeks prior to enrollment.
3. Participants who have received a live vaccine injection within 4 weeks prior to enrollment.
4. Patients with central nervous system (CNS) diseases unrelated to lymphoma central nervous system involvement (e.g., cerebral aneurysm, epilepsy, stroke, Alzheimer's disease, psychiatric disorders, etc.). Lymphoma central nervous system involvement or gastrointestinal tract involvement is not an exclusion criterion, but eligibility for enrollment shall be determined by the investigator.
5. Patients with severe active infections (except uncomplicated urinary tract infections and bacterial pharyngitis), or those currently receiving intravenous antibiotic therapy. However, prophylactic use of antibiotics, antiviral drugs, and antifungal drugs is permitted.
6. Patients who are positive for hepatitis B surface antigen (HBsAg) or positive for hepatitis B virus (HBV) DNA in peripheral blood.
7. Patients who are positive for hepatitis C virus (HCV) antibody and positive for hepatitis C virus (HCV) RNA in peripheral blood.
8. Patients with other acquired or congenital immunodeficiency diseases, including but not limited to those positive for human immunodeficiency virus (HIV) antibody; patients with cytomegalovirus (CMV) DNA test value > 400 copies/mL; patients with positive syphilis test results.
9. Patients with heart failure classified as Grade III or IV according to the New York Heart Association (NYHA) Functional Classification (see Appendix II).
10. Patients with a history of other primary malignancies, except for the following cases:Non-melanoma skin cancer (e.g., basal cell carcinoma of the skin) cured by resection;In situ carcinoma cured (e.g., cervical cancer, bladder cancer, breast cancer, etc.);Other primary malignancies with no recurrence detected for more than 5 years after treatment.
11. Patients with a history of solid organ transplantation.
12. Patients with a history of autoimmune diseases (predominantly characterized by abnormal cellular immunity), as well as patients with immunodeficiency or those requiring immunosuppressive therapy.
13. Patients who received investigational drugs from other interventional clinical trials within 3 months prior to signing the Informed Consent Form (ICF).
14. Pregnant women or women who are breastfeeding.
15. Patients with psychiatric disorders, consciousness disturbances, or central nervous system (CNS) diseases.
16. Patients whose toxic effects from prior treatment have not resolved to baseline or ≤ Grade 2 (per NCI-CTCAE Version 5.0, alopecia excluded).
17. Medication use:Corticosteroids: Use of therapeutic-dose corticosteroids within 72 hours prior to CAR-T cell infusion; however, physiological-dose corticosteroid replacement is permitted (hydrocortisone < 12 mg/m²/day or its equivalent dose)；Systemic antineoplastic therapy: Failure to discontinue systemic antineoplastic therapy for at least 2 weeks or 5 drug half-lives prior to T cell apheresis (except for BTK inhibitors in patients with CLL); the interval between T cell apheresis and the use of immune checkpoint inhibitors is less than 3 drug half-lives.
18. Patients with active pulmonary infections.
19. Patients with contraindications to peripheral blood apheresis.
20. Patients deemed unsuitable for participation in this trial by the investigator after careful consideration for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-29 (Estimated); Primary Completion 2029-11-28 (Estimated); Study Completion 2029-11-28 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Safety of BAFF-R Chimeric Antigen Receptor T-Cell Injection (BAFF-R CAR-T) in Subjects with Relapsed and Refractory BAFF-R-Positive B-Cell Lymphoma, and Exploration of the Maximum Tolerated Dose (MTD) | Day 28 after treatment
  The possible adverse reactions recorded in each item were evaluated. The highest dose at which fewer than 2 out of 6 subjects (i.e., < 2/6) experience Dose-Limiting Toxicity (DLT) (with at least 6 subjects in this dose group having received BAFF-R CAR-T infusion and completed the DLT observation period).

SECONDARY OUTCOMES:
Objective response rates (ORR) | Day 28, Month 2, Month 3, Month 6, Month 12 ,Month 24 after treatment
Overall survival (OS) | Day 28, Month 2, Month 3, Month 6, Month 12 ,Month 24 after treatment
Progression-free survival (PFS) | Day 28, Month 2, Month 3, Month 6, Month 12,Month 24 after treatment
Complete remission rate (CRR) | Day 28, Month 2, Month 3, Month 6, Month 12,Month 24 after treatment
Pharmacokinetics - Cmax | Day 28, Month 2, Month 3, Month 6, Month 12 ,Month 24 after treatment
  The maximum transgene level at Tmax
Total B Cells (CD19+ B Cells) Absolute Count | Day 28, Month 2, Month 3, Month 6, Month 12，Month 24 after treatment
  Evaluate the overall depletion efficiency of B cells by CAR-T
Pharmacokinetics - Tmax | Day 28, Month 2, Month 3, Month 6, Month 12 ,Month 24 after treatment
  Time to peak transgene level
Pharmacokinetics - AUC0-28days | Day 28, Month 2, Month 3, Month 6, Month 12 ,Month 24 after treatment
  Area under the curve of CAR T cells from time zero to Day 28